CLINICAL TRIAL: NCT05571449
Title: Efficacy of the Use of 3D Printing Models in the Treatment of Tibial Plateau Fractures: a Prospective Randomized Clinical Trial
Brief Title: Efficacy of the Use of 3D Printing Models in the Treatment of Tibial Plateau Fractures: a Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro-José Torrijos-Garrido (Other)
Responsible Party: Sponsor-Investigator, Pedro-José Torrijos-Garrido, Principal Investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIBIA3D
Record Dates: First submitted 2022-09-29; First posted 2022-10-07 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Tibial Plateau Fracture
Keywords: 3D printing; Tibial fracture
MeSH Terms: conditions — Tibial Plateau Fractures; Tibial Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Planning of tibial plateau fracture osteosynthesis by using a three-dimensional model of the fracture.
  Interventions: Procedure: Open reduction and internal fixation; Procedure: Standard osteosynthesis planning; Procedure: 3-D model osteosynthesis planning
- Control group (Other): Standard planning of tibial plateau fracture osteosynthesis (by plain radiography and computed tomography imaging).
  Interventions: Procedure: Open reduction and internal fixation; Procedure: Standard osteosynthesis planning

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Internal fixation of the fracture
Procedure: Standard osteosynthesis planning — Plain radiograph and CT images are used
Procedure: 3-D model osteosynthesis planning — A 3D plastic model made from CT images is used
  Arms: Experimental group

SUMMARY:
TIBIA3D is a randomized, open and prospective clinical trail that evaluates the use of preoperative 3D printing in the surgical treatment of patients with tibial plateau fractures

DETAILED DESCRIPTION:
Randomized, open and prospective study.

Once the surgical indication for osteosynthesis has been established after having suffered a tibial plateau fracture, the patients will be randomized in a 1:1 ratio to one of the tfollowing treatment groups:

Control group: images obtained by plain radiography and computed tomography are used in the planning of osteosynthesis of the tibial plateau fracture.

Experimental group: in the planning of tibial plateau fracture osteosynthesis, in addition to images obtained by plain radiography and computed tomography, a three-dimensional plastic model printed by processing the tomography images is used.

Patients (or their legal representatives) must sign the consent before randomization.

After surgery, a follow-up will be carried out at 3, 6 and 12 months, visits in which data will be collected regarding the physical examination, radiological examination, pain and questionnaires will be filled out regarding the functionality of the knee and perception of health status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tibial plateau fracture requiring surgical treatment.
* Age equal to or greater than 18 years.
* Signature of informed consent in writing according to current legislation before collecting any information.

Exclusion Criteria:

* Pregnancy in progress.
* Presence of serious systemic pathology or another situation that contraindicates treatment
* Presence of other fractures in the ipsilateral femur or tibia that condition the surgical treatment of the tibial plateau fracture.
* Findings in the physical examination, in the results of the tests or other medical, social or psychopathological factors that, in the opinion of the investigators, could negatively influence the study.
* Inability to grant informed consent in the absence of a legal representative.
* Inability to follow instructions or collaborate during the development of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Surgical time | Week 1
  Surgical time will include the time from skin incision to wound closure
Fluoroscopy time. | Week 1
  Intraoperative fluoroscopy time will be counted after incision and before wound closure.

SECONDARY OUTCOMES:
Ease of surgical planning with 3d printing | Week 1
  Form filled out by the surgeon before the intervention to find out if the three-dimensional impression of the fracture has changed from the original preoperative planning that it had previously
Complications | Week 1 - 12 months
  The incidence of complications, such as superficial wound infection, deep wound infection, iatrogenic neurological symptoms, reduction loss and fixation failure, will be recorded in both groups.

OTHER OUTCOMES:
Visual Analogis Scale for Pain | 6 weeks - 12 months
  VAS measure the intensity of the pain that the patient describes. It consists of a horizontal line of 10 centimeters, with 0cm being "no pain" and 10cm being "extreme pain".
KOOS Questionarie | 6 weeks - 12 months
  The Knee injury and Osteoarthritis Outcome Score (KOOS) has been developed as an instrument to assess the patient's opinion about their knee and associated problems It has to separate sections ("Knee Score" and "Functional Score") that are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
EuroQol-5D Questionarie | 6 weeks - 12 months
  Generic instrument for measuring health-related quality of life, in which the individual himself assesses his health status (0-100 score)
WOMAC Questionarie | 6 weeks - 12 months
  It is the most widely used questionnaire to assess the results after knee and hip arthroplasty in patients with osteoarthritis in the lower extremity (0-68 score)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Torrijos Garrido, MD, PhD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (1):
- Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No